CLINICAL TRIAL: NCT03223402
Title: NEVIRAPINE Plus LAMIVUDINE (3TC) for HIV Maintenance Therapy - A Single Center Pilot Study
Brief Title: Nevirapine + 3TC Based Maintenance Therapy for HIV Infection
Acronym: NVP+3TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, pietro vernazza, Chief Div. Infectious Diseases, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BASEC Nr. 2016-01963
Record Dates: First submitted 2016-12-15; First posted 2017-07-21 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Lamivudine

STUDY DESIGN:
Intervention Model Description: Pilot study, one arm. We do not evaluate a specific drug. It is an Evaluation of a combination with just two instead of three drugs for the Treatment of HIV
Oversight: Data Monitoring Committee: No

ARMS (1):
- nevirapine plus lamivudine (Experimental): patients from one Center switching from a Nevirapine based Regimen on Nevirapine + 3TC
  Interventions: Other: Nevirapine plus lamivudine

INTERVENTIONS:
Other: Nevirapine plus lamivudine — In this Pilot study, the efficacy of a bi-therapy consisting of NVP+3TC instead of NVP+2NRTI should be evaluated before a large multicenter study evaluating this combination is started.

SUMMARY:
Type of study: Investigator initiated clinical study Study design: One arm, open label, pilot study (n=10) Research question Is treatment with Nevirapine + 3TC sufficient for HIV maintenance Risk Category B (no investigational drugs, non standard Tx) Therapies with 2 drugs are often done in HIV-maintenance. This is a systematical evaluation of such a two drug trial. Rescue therapy is well defined within the protocol. Centers (n) St. Gallen only Participants 10 HIV Patients already on nevirapine + 2 non-nuke RT-Inhibitors Study duration 24 weeks primary observation period after study termination, patients may opt to continue on the bi-therapy. Clinical follow up will then continue Sponsor/Investigator Pietro Vernazza, Kantonsspital St. Gallen Principal investigator Pietro Vernazza, MD. Kantonsspital St. Gallen Co-Investigators Patrick Schmid, MD, Matthias Hoffmann, MD

Financial source None (Pilot Study) If study demonstrates good results, an SNF grant proposal will be submitted

DETAILED DESCRIPTION:
This is a pilot study to evaluate the efficacy of a two drug combination for Long term HIV maintenance therapy.

The study is conducted in order to confirm the feasibility of the combination of Nevirapine and lamivudine (3TC) in patients with long term fully suppressive therapy.

Patients (n=10) with a stable (>6 months) Nevirapine based triple therapy and a full viral load suppression for at least 2 years will continue their therapy for 6 months with Nevirapine+3TC.

The primary endpoint is treatment failure defined as an HIV-RNA value >100 cp/ml, confirmed by a second measurement.

Preliminary stopping rules are defined if results indicate futility. Futility is defined as a situation, where the investigators would stop their plan to conduct a multicenter comparative trial. Futility is reached, when the study documents more than 1 failure in the first 5 patients over 24 weeks of observation or more than 2 failures in all 10 patients.

Only 10 patients will be followed in this single center pilot study.

After an amendement (April 2017) the total number of 20 patients was increased to 20. Futility was defined as more than 2 failures in 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV-pos, 18 years
* Stable ART, Nevirapine based (plus 2 nukleotide-analogues), at least 6 months
* Viral load suppression at least 24 months Prior to inclusion (<50cp/ml)

Exclusion Criteria:

* chronic Hepatitis B necessitating tenofovir therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure defined as HIV-RNA > 100 cp/ml | 24 weeks
  Patients reaching a viral load measurement >100cp /ml (confirmed) within the first 24 weeks of therapy with monthly HIV-RNA testing.

CONTACTS AND LOCATIONS:
Overall Officials: Pietro L Vernazza, MD, Principal Investigator — KSSG
Locations (1):
- Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No
not planned